CLINICAL TRIAL: NCT06592274
Title: A Multicenter, Randomized, Double-blind Phase 2 Clinical Study Evaluating the Efficacy and Safety of Different Administration Regimens of HB0017 Injection in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: A Phase 2 Study of HB0017 in Psoriasis Patients
Acronym: HB0017
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HB0017-PsO-02-02
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis (PsO)
Keywords: HB0017; psoriasis; longer dose regimen
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Group 1 (Experimental): HB0017 higer dose plus longer dose regimen
  Interventions: Biological: HB0017
- Experimental Group 2 (Experimental): HB0017 higer dose plus shorter dose regimen
  Interventions: Biological: HB0017
- Experimental Group 3 (Experimental): HB0017 low dose plus shortest dose regimen
  Interventions: Biological: HB0017

INTERVENTIONS:
Biological: HB0017 — 300mg Q12W
  Arms: Experimental Group 1
Biological: HB0017 — 300mg Q8W
  Arms: Experimental Group 2
Biological: HB0017 — 150mg Q4W
  Arms: Experimental Group 3

SUMMARY:
This study is a randomized, double-blind phase 2 clinical trial aimed at exploring the efficacy, safety, and immunogenicity of HB0017 injection with different dosing regimens in the treatment of moderate to severe plaque psoriasis in subjects

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-75 years (inclusive)
* Chronic plaque psoriasis (PSO) for at least 6 months prior to the randomization.
* Psoriasis Area Severity Index (PASI) >=12 and body surface area (BSA) affected by PSO >=10% and Static Physician Global Assessment (sPGA) score >=3.
* Subjects who are suitable for systemic treatment or phototherapy for psoriasis as judged by the investigator
* Subjects who are able to use effective contraception from the screening period to 6 months after the last dose

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and/or guttate psoriasis) at screening or baseline Drug-induced psoriasis
* Ongoing use of prohibited treatments
* Any active infection (other than common cold) within 14 days
* Serious infection defined as requiring hospitalization or iv anti-infective(s) within 1 month prior to randomization
* Have previously received any drug that directly targets IL-17 or IL-17 receptor
* Have concurrent or recent use of any biologic agent within the following washout periods: etanercept <28 days; infliximab and adalimumab <60 days; golimumab < 90 days; anti-IL-12/anti-IL-23 or anti-IL-23p19 antibody drugs <6 months; or other anti-psoriatic therapy not listed herein within its 5 half-lives prior to randomization
* A history of inflammatory bowel disease or other serious autoimmune disease
* Previously diagnosed with serious mental illness such as anxiety, depression or suicidal tendency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving PASI 90 response | Week 12
  The PASI75 response assessments are based on at least 90% improvement in PASI score from Baseline.
Proportion of subjects achieving sPGA 0/1 | Week 12
  The sPGA is a physician's determination of the participant's psoriasis lesions overall at a given time point categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's psoriasis is assessed as clear (0), Almost clear (1), mild (2), moderate (3), severe (4). An sPGA 0/1 response was defined as a post-baseline sPGA score of 0 or 1.

SECONDARY OUTCOMES:
Proportion of subjects achieving PASI 75 response | Week 12
  The PASI75 response assessments are based on at least 75% improvement in PASI score from Baseline.
Proportion of subjects achieving PASI 100 response | Week 12
  The PASI100 response assessments are based on 100% improvement in PASI score from Baseline
PASI 90 response maintainance at week 48 | Week12-48
  Proportion of subjects maintaining PASI 90 response at Week 48 among those with PASI 90 response at Week 12
sPGA 0/1 response maintainance at week 48 | Week12-48
  Proportion of subjects maintaining sPGA 0/1 response at Week 48 among those with sPGA 0/1 response at Week 12.

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Southern Medical University Dermatology Hospital, Guangzhou, Guangdong
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - Jiangsu University Affiliated Hospital, Zhenjiang, Jiangsu
  - Jilin University Second Hospital, Changchun, Jilin
  - Shandong First Medical University Affiliated Dermatology Hospital, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Xingtai People's Hospital, Xingtai, Shandong
  - Shanxi Medical University Second Hospital, Taiyuan, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jiaxing First Hospital, Jiaxing, Zhejiang
  - Wenzhou Medical University Affiliated First Hospital, Wenzhou, Zhejiang
  - Guangdong Provincial People's Hospital, Guangzhou
  - Ningbo Second Hospital, Ningbo

IPD SHARING:
Plan to Share IPD: No